CLINICAL TRIAL: NCT05355324
Title: Anemia is a Risk Factor for Readmission and Death of Lower Respiratory Infections in Older Adults
Brief Title: Risk Factor for Readmission and Death of Lower Respiratory Infections in Older Adults
Status: Completed | Type: Observational
Sponsor: Beijing Tongren Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: YuHe_1987
Record Dates: First submitted 2022-04-21; First posted 2022-05-02 (Actual); Last update posted 2022-05-02 (Actual); Status verified 2022-04

CONDITIONS: Lower Respiratory Infection; Anemia; Readmission; Death
MeSH Terms: conditions — Anemia; Death

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- anemia: patients with anemia
  Interventions: Other: no intervention
- non-anemia: patients without anemia
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — no intervention

SUMMARY:
Lower respiratory tract infection(LRTI) is a prevalent disease that threatens the health of older people worldwide. Anemia is also a common disorder in the elderly, and its prevalence increases significantly with age. Most factors that contribute to the development of anemia are improvable. Therefore, we investigated whether anemia was a risk factor for LRTI-caused readmission and death in the elderly occurring within 1 year of discharge from the hospital.

DETAILED DESCRIPTION:
Objectives: To investigate the effect of anemia on readmission and deaths in the older adults following lower respiratory tract infection (LRTI)-caused hospitalization.

Design: A retrospective cohort study. Setting and Participants: Older patients (age: ≥ 80 years) hospitalized at the Department of Geriatrics, from March 2016 to December 2019 to undergo treatment for LRTIs were included.

Methods: The patients were divided into two groups (anemia and non-anemia) based on the level of hemoglobin. They were kept under observation till the occurrence of mortality event or 1 year after discharge. The primary follow-up outcome was LRTI-caused readmission and/or death.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 80 years
* lower respiratory tract infection

Exclusion Criteria:

* Died at the time of first admission
* Active malignancy
* Tuberculosis
* Anemia caused by gastrointestinal bleeding of unknown origin
* Achalasia of the cardia
* Could not be followed up after discharge
* Data were missing

Ages: 80 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Elderly patients (age: ≥ 80 years), hospitalized (from 31 March 2016 to 27 December 2019) at the Department of Geriatrics of a hospital in Beijing, China, and were with lower respiratory tract infection(LRTI) (including pneumonia and acute exacerbation of chronic obstructive pulmonary disease) were included. 215 patients (age: >/=80 years) who were hospitalized due to LRTI and discharged after being cured were studied. Of these 215 patients, 149 belonged to the anemia group, and 66 belonged to the non-anemia group. The mean age of the cohort at the time of inclusion was 88.73 (SD 4.765) years, and 77.2% of the patients were men.
Sampling Method: Non-Probability Sample
Enrollment: 215 (Actual)
Dates: Start 2016-03-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Number of Patients with Readmission and/ or Death Caused by Lower Respiratory Tract Infection(LRTI) within One Year of Discharge | March 2016 to 27 December 2019
  Number of Patients with Readmission Caused by LRTI within One Year of Discharge. Number of Patients with Death Caused by LRTI within One Year of Discharge.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] He Y, Chen Y, Cao K, Zheng H. Effect of Anemia on Readmission and Death in Octogenarian Patients with Lower Respiratory Tract Infections: A Retrospective Cohort Study. Int J Clin Pract. 2022 Oct 27;2022:4566936. doi: 10.1155/2022/4566936. eCollection 2022. PMID 36349057